CLINICAL TRIAL: NCT05013060
Title: An Assessment of the Efficacy of Microencapsulated Sodium Butyrate and a Probiotic Mixture in Patients With Irritable Bowel Syndrome - a Randomized Double-blind Placebo-controlled Study
Brief Title: The Efficacy of Sodium Butyrate and Probiotics in Patients With Irritable Bowel Syndrome
Acronym: IBS-Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Biotic Sp. z o.o. (Industry)
Collaborators: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Anita Gąsiorowska, MD, PhD, Nordic Biotic Sp. z o.o.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT/NB/110/2019/PR-MS-PS
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Probiotics; Butyric acid; Microencapsulated sodium butyrate
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The mixture of probiotics and microcapsulated sodium butyrate (Active Comparator): One billion of the following strains: Bifidobacterium lactis FloraActive 32269, Bifidobacterium longum FloraActive 32946, Bifidobacterium bifidum FloraActive 32043, Lactobacillus rhamnosus FloraActive 19070-2, Lactobacillus acidophilus FloraActive 32418 and 150 mg microcapsulated sodium butyrate, and 64 mg fructooligosaccharides
  Interventions: Dietary Supplement: Probiotics and microcapsulated sodium butyrate
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotics and microcapsulated sodium butyrate — The patients who give their consent to take part in this study, will receive an oral microencapsulated sodium butyrate and a mixture of probiotics formulation 2 times a day for a period of 12 weeks.
  Arms: The mixture of probiotics and microcapsulated sodium butyrate
Dietary Supplement: Maltodextrin — The patients who give their consent to take part in this study will receive an oral maltodextrin as placebo 2 times a day for a period of 12 weeks.
  Arms: Placebo

SUMMARY:
According to current IBS management guidelines, probiotic administration reduces IBS-associated symptoms and improves the quality of life. The purpose of this study is to assess the effects of the combined formulation comprising microencapsulated sodium butyrate and a probiotic mixture of two Lactobacillus strains (L. rhamnosus and L. acidophilus) and three Bifidobacterium strains (B. longum, B. bifidum, and B. lactis) on the incidence and severity of clinical symptoms in patients diagnosed with irritable bowel syndrome (IBS) based on the Rome IV criteria.

Microencapsulated sodium butyrate is a short-chain fatty acid (SCFA) with biological effects on the gastrointestinal mucosa; it constitutes a key source of energy for enterocytes. Butyrate was shown to have a trophic effect on the colon epithelium and to help restore the disrupted structural and functional integrity of the gastrointestinal tract. These unique properties of sodium butyrate result in its beneficial effects on the abdominal symptoms (such as diarrhea, constipation, abdominal pain) in patients with IBS. This study will assess the effects of the mixture of sodium butyrate and multi-strain probiotic on the rate and severity of clinical symptoms in IBS patients, by taking into account their nutritional status and body composition.

DETAILED DESCRIPTION:
The study schedule includes five visits:the screening/baseline visit, whose purpose is to qualify patients to be included in the study, the randomization visit (visit 0), at which patients will be given a probiotic/butyric acid or placebo, and three follow-up visits (at weeks 4, 8, and 12 after randomization).

All patients will undergo:

1. A physical examination - at each visit;
2. Nutritional status assessment - at visit 0 and at weeks 4 and 12 of treatment;
3. Anthropometric measurements - at visit 0 and at weeks 4 and 12 of treatment;
4. Body composition analysis via bioelectrical impedance analysis (BIA) with the use of a Bodystat machine - at visit 0 and at 4 and 12 weeks of treatment;
5. Laboratory tests (including complete blood count; liver function tests; bilirubin, amylase, creatinine, CRP, and glucose levels; electrolytes; and an SARS-CoV2 antigen cassette test conducted by a doctor) at the screening visit; and cytokines (IL-6 and macrophage inflammatory protein 1β (MIP-1ß)) at visit 0 and at weeks 4 and 12 of treatment;
6. Disease severity will be rated with the IBS symptom severity score (IBS-SSS) developed by Francis, Morris, and Whorwell, with mild, moderate, and severe cases indicated by scores of <175, 175-300, and >300, respectively. In addition, the following scales will be used to assess IBS treatment efficacy: IBS-Quality of Life (IBS-QOL), IBS-Global Improvement Scale (IBS-GIS), and IBS - Adequate Relief (IBS-AR).
7. The number and type of bowel movements will be assessed with the Bristol Stool Formation scale.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged from 18 to 70 years, inclusive;
2. Good physical and mental condition assessed based on the patient's history and physical examination;
3. Laboratory test results (complete blood count, blood chemistry panel) within normal limits or considered not to be clinically significant by the Investigator; negative SARS-CoV-2 antibody test;
4. A voluntarily provided written informed consent;
5. Diagnosis of IBS based on the Rome IV criteria, e.g. recurrent abdominal pain at least one day a week for the last three months, associated with two or more of the following symptoms (these should be present for the last three months, with the onset of symptoms six months before diagnosis):

   * related to defecation
   * associated with a change in stool frequency and/or
   * associated with a change in stool form (appearance)

   Patients with any of the following forms of IBS will be included:
   * IBS-D - more than 25% of BSF type 6 and 7 stools, and less than 25% of type 1 and 2 stools.
   * IBS-C - more than 25% of BSF type 1 and 2 stools, with less than 25% of type 6 and 7 stools.
   * IBS-M - more than 25% of BSF type 6 and 7 stools and also more than 25% of type 1 and 2 stools.
   * at least moderate symptom severity defined as an IBS-SSS score of >175 (5 items, maximum score 500).
6. The following medications are allowed during this study, provided they have been used at a stable dose and for at least 1 month prior to the study:

   1. contraceptive pills or intramuscular contraceptives,
   2. hormone replacement therapy (estrogen/progesterone),
   3. L-thyroxine,
   4. antidepressants at low doses (up to 25 mg of amitriptyline, nortriptyline, or selective serotonin reuptake inhibitor per day)
   5. antihypertensives at low doses (diuretics, angiotensin converting enzyme inhibitors angiotensin receptor antagonists).

Exclusion Criteria:

1. Unclassified IBS;
2. Cardiovascular disorders: uncontrolled hypertension (blood pressure >170/100 mmHg), cerebrovascular disease;
3. Respiratory disorders (asthma, chronic obstructive pulmonary disease [COPD]).
4. Hepatic impairment (including status post cholecystectomy), renal impairment, and unexplained blood biochemistry abnormalities: serum creatinine levels over twice the upper limit of normal, AST or ALT levels over twice the upper limit of normal.
5. Gastrointestinal conditions other than IBS, including clinical or endoscopic diagnosis of gastroenteritis.
6. Endocrine disorders, including diabetes mellitus (fasting blood glucose >11 mmol/L) and elevated TSH levels.
7. Severe neurological conditions, with psychosis;
8. Malignancy;
9. Pregnancy or breastfeeding;
10. Hypersensitivity to soy;
11. Lactose intolerance;
12. The use of gastrointestinal motility stimulants or dietary fiber supplements during the 2 weeks preceding the clinical study;
13. The use of antithrombotic drugs;
14. A surgical procedure scheduled during the course of the clinical study;
15. Current probiotic use and refusal to undergo a 3-month washout period;
16. Antibiotic therapy during the 3 months preceding the study;
17. Antibiotic use during the study;
18. Being included in another clinical study during the previous 3 months;
19. History of alcohol or substance;
20. Inability to strictly adhere to the Investigators' instructions regarding study procedures and protocol requirements.abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in severity of IBS symptoms using IBS Severity Scoring System (IBS-SSS) | Severity of symptoms from baseline at 4, 8 and 12 weeks of intervention
  IBS-SSS is a 5-question survey that asks: 1. the severity of abdominal pain, 2. frequency of abdominal pain, 3. severity of abdominal distention, 4.dissatisfaction with bowel habit, and 5. interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Each of the five question generates a maximum score of 100 point, and total scores can range from 0-500 with higher scores indicating severe symptoms.
Improvement or worsening of IBS global symptoms using Global Improvement Scale (IBS-GIS) | Improvement/worsening assessed after 4, 8 and 12 weeks of intervention
  IBS-Global Improvement Scale asseses IBS symptoms using a patient-defined 7 point Linkert scale ranging from symptoms substantially worse to substantially improved.
  Patients answer the question "Have you felt any change in the severity of your symptoms over the past 7 days compared to how you felt before the medicine was given?
  The answers are recorded based on the 7-point scale:
  1. = I feel that the symptoms have worsened significantly
  2. = I feel that the symptoms have moderately worsened
  3. = I feel that the symptoms have slightly worsened
  4. = I feel no change
  5. = I feel a slight improvement
  6. = I feel moderate improvement
  7. = I feel significant improvement IBS-GIS score indicates: improvement if is >4 or worsening if is<4, no change if is 4.
Changes in an adequate relief | Adequate Relief after 4, 8 and 12 weeks of interventions
  IBS-Adequate Relief (IBS-AR) is a dichotomous single item that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms? The answer is YES or NO.
Changes in Quality of Life | Quality of Life from baseline at 4, 8 and 12 weeks of intervention
  The IBS-Quality of Life (IBS-QOL) is a 34-item measure assessing the degree to which IBS interferes with patient quality of life. Each item is rated on a 5-point Likert scale, thus yielding a total score that has a theoretical range of 34 to 170, with higher scores indicating worse QOL.

SECONDARY OUTCOMES:
Changes in number and type of stools | From baseline for 12 weeks of intervention in 1 week intervals
  Number of stools per day and type of stools assessed before intervention and then 3 times a week. Type of stools assessed using the Bristol Stool Formation Scale. Bristol Scale is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea.
Changes in severity of pain | From baseline for 12 weeks of intervention in 1 week intervals
  The severity of pain assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no pain, and 1-4 the severity of pain with higher scores indicating worse pain.
Changes in flatulence/abdominal distension | From baseline for 12 weeks of intervention in 1 week intervals
  The severity of flatulence/abdominal distension assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no flatulence/abdominal distension, and 1-4 the severity of flatulence/abdominal distension with higher scores indicating worse flatulence/abdominal distension.
Changes in Body Mass Index (BMI) | From baseline at 4 and 12 weeks of intervention
  The effect of intervention on the patient's weight
Body composition analysis | From baseline at 4 and 12 weeks of intervention
  Body composition will be measured via bioelectrical impedance analysis with the use of a Bodystat machine.

OTHER OUTCOMES:
Changes in interleukin 6 (IL-6) and macrophage inflammatory protein 1β (MIP-1ß) levels | From baseline at 4 and 12 weeks of intervention
  IL-6 and MIP-1ß levels will be measured in the sera of patients using commercially available immunoenzymatic tests.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Gąsiorowska, MD, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Lodz, Poland

REFERENCES:
- [Derived] Gasiorowska A, Romanowski M, Walecka-Kapica E, Kaczka A, Chojnacki C, Padysz M, Siedlecka M, Bierla JB, Steinert RE, Cukrowska B. Effects of Microencapsulated Sodium Butyrate, Probiotics and Short Chain Fructooligosaccharides in Patients with Irritable Bowel Syndrome: A Study Protocol of a Randomized Double-Blind Placebo-Controlled Trial. J Clin Med. 2022 Nov 7;11(21):6587. doi: 10.3390/jcm11216587. PMID 36362815